CLINICAL TRIAL: NCT00576810
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 4 Weeks Treatment With Sodium Picosulfate [Dulcolax®, Laxoberal®]Drops 10 mg Administered Orally, Once Daily, in Patients With Functional Constipation
Brief Title: Sodium Picosulphate vs. Placebo in Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1062.7; EURDRACT2007-002087-10
Record Dates: First submitted 2007-10-29; First posted 2007-12-19 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — picosulfate sodium

INTERVENTIONS:
Drug: sodium picosulphate

SUMMARY:
The objective ot the study is to compare the efficacy and safety of 4 weeks treatment with sodium picosulphate drops 10mg to placebo in patients with functional constipation. In addition the effect of treatment on quality of life and general health status will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged 18 and above
2. Suffering from functional constipation, according to their medical history, as defined by the Rome III diagnostic criteria Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.

   1. Must include 2 or more of the following:

      * straining during at least 25% of the defecations
      * lumpy or hard stools in at least 25% of the defecations
      * sensation of incomplete evacuation for at least 25% of the defecations
      * sensation of anorectal obstruction/blockade for at least 25% of the defecations
      * manual manoeuvres to facilitate at least 25% of the defecations (e.g. digital evacuation, support of the pelvic floor)
      * fewer than 3 defecations per week
   2. Loose stools are rarely present without the use of laxatives
   3. There are insufficient criteria for irritable bowel syndrome (IBS) (i.e. recurrent abdominal pain or discomfort is not the predominant symptom associated with defecation or a change in bowel habit, and with features of disordered defecation)
3. Able and willing to complete a daily e-diary
4. Able and willing to use the trial rescue medication (i.e. 10 mg bisacodyl suppositories)
5. Signed and dated written informed consent prior to enrolment into the study in accordance with GCP and local legislation

Exclusion Criteria:

1. Eating disorders such as anorexia nervosa and bulimia, as a cause of excessive use of laxatives
2. Patients whose constipation is caused by primary organic disease of the colon or pelvic floor
3. Patients with metabolic disorders, neurological disorders, severe or psychiatric disorders, or any other significant disease or intercurrent illness (e.g. abdominal/gastrointestinal surgery) that, in the Investigators opinion, would interfere with participation in the trial
4. Patients with restricted mobility (e.g. wheelchair bound, or bed-ridden) that, in the Investigators opinion, would interfere with participation in the trial
5. Patients with a known hypersensitivity to sodium picosulphate, bisacodyl or any other ingredient in the study medication (sodium picosulphate and matching placebo drops, bisacodyl suppositories)
6. Patients with ileus, intestinal obstruction, acute surgical abdominal conditions (such as acute appendicitis and acute inflammatory bowel diseases), or severe dehydration
7. Patients with anal fissures or ulcerative proctitis with mucosal damage
8. Patients with known clinically significant abnormal electrolyte values
9. Patients whose concomitant therapy includes an opioid medication (e.g. morphine, codeine)
10. Constipation which, in the Investigators opinion, is caused by medication (e.g. anticholinergics)
11. Patients who are not willing to discontinue the use of prohibited concomitant therapy (see Section 4.2.2)
12. Pre-menopausal women (last menstruation £ 1 year prior to signing informed consent) who:are nursing (breast-feeding) or who are pregnant OR who are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study.
13. Participating in another trial with an investigational product with 1 month of enrolment into this study
14. Drug or alcohol abuse
15. Concomitant use of antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this trial is the mean number of complete spontaneous bowel movements (CSBMs) per week, during the 4 week treatment phase of the trial. | 4 weeks

SECONDARY OUTCOMES:
Number of CSBMs per week, at each weekly time point during the treatment phase of the trial (i.e. at each of weeks 1, 2, 3 and 4) | 4 weeks
Number of spontaneous bowel movements (SBMs) per week after the first intake of the study medication | 4 weeks
Time to first SBM following the first intake of the study medication | 4 weeks
Number of patients with an increase of ≥ 1 CSBM per week compared with the last 7 days of the baseline period | 4 weeks
Number of patients with ≥ 1 CSBM a day | 4 weeks
Number of patients with ≥ 3 CSBMs per week | 4 weeks
Number of premature withdrawals | 4 weeks
Number of patients who have used rescue medication | 4 weeks
Change from baseline in mean score per week for constipation symptoms | 4 weeks
Change from baseline in the patients' score per week for overall satisfaction with bowel habits and bothersomeness of constipation symptoms | 4 weeks
Final global assessment of efficacy by the investigator (good, satisfactory, not satisfactory, bad) | 4 weeks
Final global assessment of efficacy by the patient (good, satisfactory, not satisfactory, bad) | 4 weeks
Quality of Life (SF-36v2and PAC-QOL) | 4 weeks
Blood pressure | 4 weeks
Number of participants with abnormal serum electrolyte laboratory parameters | 4 weeks
Number of participants with abnormal serum chemistry laboratory parameters | 4 weeks
Final global assessment of tolerability by the investigator (good, satisfactory, not satisfactory, bad) | 4 weeks
Final global assessment of tolerability by the patient (good, satisfactory, not satisfactory, bad) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (43):
- Germany (43):
  - 1062.7.4926 Boehringer Ingelheim Investigational Site, Amberg
  - 1062.7.4918 Boehringer Ingelheim Investigational Site, Bad Essen
  - 1062.7.4946 Boehringer Ingelheim Investigational Site, Bergkamen
  - 1062.7.4904 Boehringer Ingelheim Investigational Site, Berlin
  - 1062.7.4929 Boehringer Ingelheim Investigational Site, Berlin
  - 1062.7.4902 Boehringer Ingelheim Investigational Site, Blankenhain
  - 1062.7.4927 Boehringer Ingelheim Investigational Site, Dortmund
  - 1062.7.4954 Boehringer Ingelheim Investigational Site, Dortmund
  - 1062.7.4949 Boehringer Ingelheim Investigational Site, Dresden
  - 1062.7.4950 Boehringer Ingelheim Investigational Site, Einbeck
  - 1062.7.4909 Boehringer Ingelheim Investigational Site, Freising
  - 1062.7.4923 Boehringer Ingelheim Investigational Site, Fürth
  - 1062.7.4912 Boehringer Ingelheim Investigational Site, Hagen
  - 1062.7.4953 Boehringer Ingelheim Investigational Site, Hamburg
  - 1062.7.4910 Boehringer Ingelheim Investigational Site, Hanover
  - 1062.7.4920 Boehringer Ingelheim Investigational Site, Herne
  - 1062.7.4944 Boehringer Ingelheim Investigational Site, Ingelheim
  - 1062.7.4936 Boehringer Ingelheim Investigational Site, Jena
  - 1062.7.4925 Boehringer Ingelheim Investigational Site, Leipzig
  - 1062.7.4931 Boehringer Ingelheim Investigational Site, Leipzig
  - 1062.7.4907 Boehringer Ingelheim Investigational Site, Leverkusen
  - 1062.7.4942 Boehringer Ingelheim Investigational Site, Ludwigsburg
  - 1062.7.4906 Boehringer Ingelheim Investigational Site, Ludwigsfelde
  - 1062.7.4941 Boehringer Ingelheim Investigational Site, Ludwigshafen
  - 1062.7.4922 Boehringer Ingelheim Investigational Site, Lüdenscheid
  - 1062.7.4930 Boehringer Ingelheim Investigational Site, Lüdenscheid
  - 1062.7.4911 Boehringer Ingelheim Investigational Site, Lützen
  - 1062.7.4916 Boehringer Ingelheim Investigational Site, Marburg
  - 1062.7.4948 Boehringer Ingelheim Investigational Site, Marl
  - 1062.7.4921 Boehringer Ingelheim Investigational Site, Oelde
  - 1062.7.4935 Boehringer Ingelheim Investigational Site, Offenbach
  - 1062.7.4903 Boehringer Ingelheim Investigational Site, Potsdam
  - 1062.7.4937 Boehringer Ingelheim Investigational Site, Recklinghausen
  - 1062.7.4956 Boehringer Ingelheim Investigational Site, Reichenbach
  - 1062.7.4905 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1062.7.4933 Boehringer Ingelheim Investigational Site, Salzkotten
  - 1062.7.4943 Boehringer Ingelheim Investigational Site, Stendal
  - 1062.7.4955 Boehringer Ingelheim Investigational Site, Stuhr
  - 1062.7.4957 Boehringer Ingelheim Investigational Site, Thedinghausen
  - 1062.7.4913 Boehringer Ingelheim Investigational Site, Wallerfing
  - 1062.7.4924 Boehringer Ingelheim Investigational Site, Wardenburg
  - 1062.7.4914 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1062.7.4901 Boehringer Ingelheim Investigational Site, Winsen